CLINICAL TRIAL: NCT03118141
Title: Cumulative Live Birth Rate With eSET After In-vitro Fertilization With Preim-plantation Genetic Screening by Next Generation Sequencing Versus Conventional In-vitro Fertilization: A Pragmatic Randomized Controlled Clinical Trial
Brief Title: Cumulative Live Birth Rate With eSET After Preimplantation Genetic Screening Versus Conventional In-vitro Fertilization
Acronym: CESE-PGS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Zi-Jiang (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Peking University Third Hospital (Other); ShangHai Ji Ai Genetics & IVF Institute (Other); RenJi Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Suzhou Municipal Hospital (Other); Renmin Hospital of Wuhan University (Other); Yantai Yuhuangding Hospital (Other); Tang-Du Hospital (Other); Nanjing Maternity and Child Health Care Hospital (Other); Guangxi Maternal and Child Health Hospital (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Guangdong Women and Children Hospital (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); Shengjing Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor-Investigator, Chen Zi-Jiang, Professor, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CESE-PGS
Record Dates: First submitted 2017-03-27; First posted 2017-04-18 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Infertility
Keywords: preimplantation genetic screening; single embryo transfer; frozen embryo transfer; cumulative live birth rate
MeSH Terms: conditions — Infertility | interventions — Base Sequence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGS group (Active Comparator): Subjects in the PGS group will have blastocyst biopsy and sequencing done with 3 good-quality embryos on Day 5. Principle of freeze-all and single thawed blastocyst transfer will be applied. The transfer order of euploid embryos will be determined by blastocyst morphologic score. The outcome of all euploids transfers within 1 year after randomization will be followed up. During study, every subject will have at most one live birth.
  Interventions: Procedure: blastocyst morphologic score; Procedure: blastocyst biopsy and sequencing; Procedure: freeze-all and single thawed blastocyst transfer
- IVF group (Active Comparator): Subjects in the IVF group will also comply with the principle of freeze-all and single thawed blastocyst transfer. The order of transfer will be determined by blastocyst morphologic score. The outcome of up to 3 transfers within 1 year after randomization will be followed up. During study, every subject will have at most one live birth.
  Interventions: Procedure: blastocyst morphologic score; Procedure: freeze-all and single thawed blastocyst transfer

INTERVENTIONS:
Procedure: blastocyst morphologic score — Blastocysts will be scored by Gardner morphologic criteria.
Procedure: blastocyst biopsy and sequencing — Three blastocysts will be biopsied on trophectoderm, sequenced with next-generation sequencing (NGS). Euploidy will transferred one by one according to morphologic score.
  Arms: PGS group
Procedure: freeze-all and single thawed blastocyst transfer — All blastocysts will be vitrified in fresh cycle. Single blastocyst will be thawed and transferred.

SUMMARY:
The purpose of this randomized clinical trial is to compare the efficacy and safety with transfer of embryos selected by next generation sequencing (NGS) versus conventional morphological criteria. Subjects with 3 or more blastocysts on day 5 of embryo culture will be randomized to the PGS or IVF group. A Freeze-all strategy and a single frozen blastocyst transfer will be performed in both PGS and IVF groups. The primary outcome is the cumulative live birth after transfers of up to 3 single blastocycsts in both groups.

DETAILED DESCRIPTION:
This is a multicenter, randomized clinical trial comparing the efficacy and safety with transfer of embryos selected by next generation sequence (NGS) and morphologic criteria versus by morphological criteria alone. Subjects who obtain 3 or more good-quality blastocysts will be randomized to PGS or IVF group. All embryos will be frozen and a single thawed blastocyst will be transferred in both PGS and IVF group. Subjects in the PGS group will have 3 blastocysts sequenced and euploid embryos will be subsequently transferred. Subjects in the IVF group will have blastocysts selected by morphology assessment. The cumulative live birth rate will be counted after transfers of all euploid embryo in the PGS group and 3 blastocysts in the IVF group within 1 year after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are participating in their first cycle of IVF or ICSI
2. Women ages 20 to 37 years.
3. Women who obtain 3 or more good-quality blastocysts defined as morphological score of inner cell mass B or A, trophectoderm C or better, and grade 4 or better on day 5 of embryo culture will be randomized.

Exclusion Criteria:

1. Women with a uterine cavity abnormality, such as a uterine congenital malformation (uterus uni-cornate, bicornate, or duplex); untreated uterine septum, adenomyosis, submucous myoma, or endo-metrial polyp(s); or with history of intrauterine adhesions.
2. Women with untreated hydrosalpinx;
3. Women who are indicated and planned to undergo PGD, for example, parental abnormal karyo-type or diagnosed with monogenic disease;
4. Women who use donated oocytes or sperm to achieve pregnancy;
5. Women with contraindication for assisted reproductive technology or for pregnancy, such as poorly controlled Type I or Type II diabetes; undiagnosed liver disease or dysfunction (based on se-rum liver enzyme testing); renal disease or abnormal serum renal function; significant anemia; history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident; uncontrolled hyper-tension, known symptomatic heart disease; history of or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma; undiagnosed vaginal bleeding.

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1215 (Estimated)
Dates: Start 2017-07-09 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate | 22 months
  Live birth is defined as the delivery of any viable infant at 28 weeks or more of gestation after our interventions, and cumulative live birth rate is calculated by dividing the number of women achieving live birth after transfers of all study-specific embryos (up to 3 transfers of single blastocycst within 1 year after randomization), by the total number of women randomized to the specific group.

SECONDARY OUTCOMES:
Rate of Good Birth Outcomes | 22 months
  Number of good birth outcomes / number of clinical pregnancies over (up to) 3 transfers within 1 year.Good Birth Outcome is defined as live birth of an infant born at ≥ 37 weeks, with a birth weight between 2500 and 4000g and without a major congenital anomaly.
Cumulative pregnancy rate | 14 months
  Number of women with clinical pregnancies over (up to) 3 transfers within 1 year / number of women randomized to the specific group. Clinical pregnancy will be diagnosed with detection of an intrauterine gestational sac.
Cumulative pregnancy loss rate | 19 months
  Number of pregnancy losses / number of clinical pregnancies over (up to) 3 transfers within 1 year.Pregnancy loss refers to a complete spontaneous abortion or a nonviable pregnancy before 28 weeks of gestation.
Multiple pregnancy rate | 22 months
  Number of multiple pregnancies / number of clinical pregnancies over (up to) 3 transfers within 1 year.
Duration of pregnancy | 22 months
  The time from the first day of last menstrual period to the day of delivery.
Birth weight | 22 months
  Weight of newborns at delivery.
Cumulative incidence of maternal and neonatal complications during whole gestation and prenatal stage | 22 months
  Number of pregnancies with complications / number of pregnancies over (up to) 3 transfers within 1 year;number of live births with neonatal complications / number of live births over (up to)3 transfers within 1 year.
Number of embryo transfers to achieve live birth | 22 months
  Number of embryo transfers the patients have gone through to achieve live birth.

OTHER OUTCOMES:
Clinical pregnancy rate after the first transfer | 4 months
  Number of women with clinical pregnancies after the first transfer / number of women randomized to the specific group.
Pregnancy loss rate after the first transfer | 9 months
  Number of pregnancy losses / number of clinical pregnancies after the first transfer .
Live birth rate after the first transfer | 12 months
  Number of women with live births after the first transfer / number of women randomized to the specific group.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dahdouh EM, Balayla J, Garcia-Velasco JA. Comprehensive chromosome screening improves embryo selection: a meta-analysis. Fertil Steril. 2015 Dec;104(6):1503-12. doi: 10.1016/j.fertnstert.2015.08.038. Epub 2015 Sep 16. PMID 26385405
- [Background] Forman EJ, Hong KH, Ferry KM, Tao X, Taylor D, Levy B, Treff NR, Scott RT Jr. In vitro fertilization with single euploid blastocyst transfer: a randomized controlled trial. Fertil Steril. 2013 Jul;100(1):100-7.e1. doi: 10.1016/j.fertnstert.2013.02.056. Epub 2013 Mar 30. PMID 23548942
- [Background] Yang Z, Liu J, Collins GS, Salem SA, Liu X, Lyle SS, Peck AC, Sills ES, Salem RD. Selection of single blastocysts for fresh transfer via standard morphology assessment alone and with array CGH for good prognosis IVF patients: results from a randomized pilot study. Mol Cytogenet. 2012 May 2;5(1):24. doi: 10.1186/1755-8166-5-24. PMID 22551456
- [Background] Scott RT Jr, Upham KM, Forman EJ, Hong KH, Scott KL, Taylor D, Tao X, Treff NR. Blastocyst biopsy with comprehensive chromosome screening and fresh embryo transfer significantly increases in vitro fertilization implantation and delivery rates: a randomized controlled trial. Fertil Steril. 2013 Sep;100(3):697-703. doi: 10.1016/j.fertnstert.2013.04.035. Epub 2013 Jun 1. PMID 23731996
- [Background] Murugappan G, Ohno MS, Lathi RB. Cost-effectiveness analysis of preimplantation genetic screening and in vitro fertilization versus expectant management in patients with unexplained recurrent pregnancy loss. Fertil Steril. 2015 May;103(5):1215-20. doi: 10.1016/j.fertnstert.2015.02.012. Epub 2015 Mar 13. PMID 25772770
- [Background] Mastenbroek S, Repping S. Preimplantation genetic screening: back to the future. Hum Reprod. 2014 Sep;29(9):1846-50. doi: 10.1093/humrep/deu163. Epub 2014 Jul 8. PMID 25006207
- [Background] Huang J, Yan L, Lu S, Zhao N, Xie XS, Qiao J. Validation of a next-generation sequencing-based protocol for 24-chromosome aneuploidy screening of blastocysts. Fertil Steril. 2016 Jun;105(6):1532-6. doi: 10.1016/j.fertnstert.2016.01.040. Epub 2016 Feb 19. PMID 26902859
- [Derived] Guo L, Guo A, Lan X, Tian S, Sun F, Su Y, Chen ZJ, Cao Y, Li Y. Oligoasthenospermia is correlated with increased preeclampsia incidence in subfertile couples undergoing in vitro fertilization and embryo transfer: a secondary analysis of a randomized clinical trial. F S Sci. 2024 Nov;5(4):386-394. doi: 10.1016/j.xfss.2024.08.003. Epub 2024 Aug 15. PMID 39153572
- [Derived] Ni T, Zhou W, Liu Y, Cui W, Liu Y, Lu J, Zhang Q, Chen ZJ, Li Y, Yan J. Excessive Exogenous Gonadotropins and Genetic and Pregnancy Outcomes After Euploidy Embryo Transfer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e244438. doi: 10.1001/jamanetworkopen.2024.4438. PMID 38564220
- [Derived] Hu M, Liu M, Tian S, Guo L, Zang Z, Chen ZJ, Li Y. Comparative analysis of pregnancy outcomes in preimplantation genetic testing for aneuploidy and conventional in vitro fertilization and embryo transfer: a stratified examination on the basis of the quantity of oocytes and blastocysts from a multicenter randomized controlled trial. Fertil Steril. 2024 Jul;122(1):121-130. doi: 10.1016/j.fertnstert.2024.02.023. Epub 2024 Feb 15. PMID 38367687
- [Derived] Yan J, Qin Y, Zhao H, Sun Y, Gong F, Li R, Sun X, Ling X, Li H, Hao C, Tan J, Yang J, Zhu Y, Liu F, Chen D, Wei D, Lu J, Ni T, Zhou W, Wu K, Gao Y, Shi Y, Lu Y, Zhang T, Wu W, Ma X, Ma H, Fu J, Zhang J, Meng Q, Zhang H, Legro RS, Chen ZJ. Live Birth with or without Preimplantation Genetic Testing for Aneuploidy. N Engl J Med. 2021 Nov 25;385(22):2047-2058. doi: 10.1056/NEJMoa2103613. PMID 34818479
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291